CLINICAL TRIAL: NCT05695430
Title: Telehealth-delivered Brief Cognitive Behavioral Therapy to Prevent Suicides in People with Physical Disabilities
Brief Title: Brief Cognitive Behavioral Therapy for People with Physical Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Lauren Khazem, Research Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021B0340
Record Dates: First submitted 2022-11-17; First posted 2023-01-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation; Disability Physical; Disability Hearing; Disability, Vision
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brief Cognitive Behavioral Therapy for People with Physical Disabilities (Experimental)
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy for People with Physical Disabilities

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy for People with Physical Disabilities — 12 sessions of of Brief Cognitive Behavioral Therapy that has been adapted for people with physical disabilities will be administered through telehelath.

SUMMARY:
The purpose of this study is to examine the effectiveness of a psychotherapy (non-medication) treatment, Brief Cognitive Behavioral Therapy for Suicide Prevention, in reducing suicide ideation and attempts for people with physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Disability impacting vision, hearing, or mobility
* Past-week suicidal ideation or past-month suicide attempt

Exclusion Criteria:

* Inability to provide informed consent
* Lack of internet connection and web camera

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Scaler for Suicide Ideation | Weekly change through treatment completion, an average of 3 months
  Past-week suicidal ideation severity

SECONDARY OUTCOMES:
Self-Injurious Thoughts and Behaviors Interview-Revised | Through treatment completion, an average of 3 months
  Suicide attempt since last assessment

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State Universitty Wexner Medical Center, Columbus, Ohio, United States